CLINICAL TRIAL: NCT03248232
Title: AssessmenTs of ThRombogenicity for trAnsCatheter aorTIc valVE Implantation by Total Thrombus-formation Analysis System (ATTRACTIVE-TTAS)
Brief Title: Assessments of Thrombus Formation in TAVI
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Kenichi Tsujita, MD, PhD, Professor of Cardiovascular Medicine, Principal Investigator, Kumamoto University
Other Study IDs: Ethics No. 1440
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases
Keywords: Transcatheter aortic valve implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is well established, and can improve clinical outcomes of patients with severe aortic valve stenosis (AS) who are inoperable or have high surgical risk. Although the rates of periprocedural bleeding events are lower in TAVI compared to those in surgical aortic valve replacement, those in TAVI still remains high. In addition, current guideline recommended the dual antiplatelet (DAPT), clopidogrel plus aspirin, for a 3- to 6-month period after TAVI, however no evidences supports this approach. The antithrombotic regimen in patients undergoing TAVI is needed to be established.

To establish the antithrombotic regimen in patients undergoing TAVI,

1. the investigators assess the changes in platelet thrombus formation and white thrombus formation in patients undergoing TAVI measured by Total Thrombus Formation Analysis System (T-TAS).
2. the investigators analyze plasma microRNAs, and shear stress by using computational fluid dynamics (CFD) to clarify the mechanistic factors regarding those changes.

ELIGIBILITY:
Inclusion Criteria:

* twenty years and older
* with the informed consent of the patient or support person in case of disability at baseline (patient intubated and ventilated)

Exclusion Criteria:

* withdrawn the informed consent
* patients with trans-apical approach
* critical illness condition (severe infectious disease, cancer, severe bleeding disorder)
* transition to the surgical AVR

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic aortic valve stenosis, undergoing transcatheter aortic valve implantation
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in T-TAS parameters (AR-chip, PL-chip) during TAVI | pre-, day 2, day 7, 1 month after device implantation
  To measure the thrombus formation area under the curve for AR-chip (AR10-AUC30), and PL-chip (PL24-AUC10) before and after TAVI.

SECONDARY OUTCOMES:
Changes in shear stress analyzed by using CFD analysis of contrast-enhanced CT | pre-, day 7 after device implantation
  To measure the shear stress of aortic valve and aorta before and after TAVI by using CFD analysis of contrast-enhanced computed tomography (CT).
Changes in von Willebrand factor multimer decrease | pre-, day 2 after device implantation
  To measure the von Willebrand factor multimer decrease by using electrophoresis
Periprocedural complication, particularly, bleeding complication defined by VARC-2 criteria. | within 30 days after device implantation

OTHER OUTCOMES:
Changes in plasma microRNAs | pre-, day 2 after device implantation
  To measure the expression of plasma microRNAs before and after TAVI by using qPCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University Hospital, Kumamoto, Japan

REFERENCES:
- [Derived] Ishii M, Kaikita K, Mitsuse T, Nakanishi N, Oimatsu Y, Yamashita T, Nagamatsu S, Tabata N, Fujisue K, Sueta D, Takashio S, Arima Y, Sakamoto K, Yamamoto E, Tsujita K. Reduction in thrombogenic activity and thrombocytopenia after transcatheter aortic valve implantation - The ATTRACTIVE-TTAS study. Int J Cardiol Heart Vasc. 2019 Mar 28;23:100346. doi: 10.1016/j.ijcha.2019.100346. eCollection 2019 Jun. PMID 30976651